CLINICAL TRIAL: NCT03225144
Title: Investigating Complex Neurodegenerative Disorders Related to Amyotrophic Lateral Sclerosis and Frontotemporal Dementia
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170131; 17-N-0131
Record Dates: First submitted 2017-07-20; First posted 2017-07-21 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-11-26

CONDITIONS: Frontotemporal Dementia; Amyotrophic Lateral Sclerosis; Progressive Supranuclear Palsy
Keywords: TDP-43; Progressive Supranuclear Palsy; Motor Neuron Disease; Frontotemporal Dementia; Corticobasal Syndrome; Natural History
MeSH Terms: conditions — Frontotemporal Dementia; Amyotrophic Lateral Sclerosis; Supranuclear Palsy, Progressive; Motor Neuron Disease; Corticobasal Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: patients who are referred with a diagnosis of frontotemporal dementia, motor neuron disorder, or related adult-onset neurodegenerative disorder to assess patient eligibility for ongoing protocols

SUMMARY:
Background:

Neurodegenerative disorders can lead to problems in movement or memory. Some can cause abnormal proteins to build up in brain cells. Researchers want to understand whether these diseases have related causes or risk factors.

Objective:

To test people with movement or thinking and memory problems to see if they are eligible for research studies.

Eligibility:

People ages 18 and older with a neurodegenerative disorder associated with accumulation of TDP-43 or Tau proteins

Design:

Participants will have a screening visit. This may take place over 2-3 days. Tests include:

Medical history

Physical exam

Questions about behavior and mood

Tests of memory, attention, concentration, and thinking

Movement measurement. The speed at which participants can stand up from a chair, tap their finger and foot, and walk a short distance will be measured. Some movements will be videotaped. They will be videotaped while they speak and read a paragraph.

Blood tests. This might include genetic testing.

Lung and breathing tests

MRI. They will lie on a table that slides into a cylinder that takes pictures of the body. Some participants will get a dye through IV.

Electromyography. A thin needle will be inserted into the muscles to measure electrical signals.

Nerve tests. Small electrodes on the skin record muscle and nerve activity.

A small piece of skin may be removed.

A skin or blood sample may be taken to create stem cells.

Optional lumbar puncture. A needle will be inserted into the space between the bones of the back to collect fluid.

If participants are not eligible for current studies, they may be contacted in the future.

DETAILED DESCRIPTION:
Objectives

The primary objective is to evaluate patients referred with a diagnosis of frontotemporal dementia (FTD), amyotrophic lateral sclerosis (ALS), or related adult-onset neurodegenerative disorders to assess patient eligibility for ongoing protocols. The secondary objective is to develop and maintain a registry of characterized patients and presymptopmatic carriers of gene mutations that cause ALS-FTD spectrum disorders. The exploratory objectives are to obtain biospecimens from clinically characterized patients to carry out laboratory-based studies aimed at understanding the molecular pathways and genetic overlap between these neurodegenerative disorders and to perform 7 tesla magnetic resonance imaging studies to identify imaging biomarkers of neurodegeneration.

Study population

Adults referred with clinical diagnoses of frontotemporal dementia, motor neuron disorder, or related adult-onset neurodegenerative disorder. Presymptomatic carriers of genes known to cause familial FTD or ALS

Design

All participants will undergo clinical tests to confirm diagnoses and to stage disease severity, including a standard battery of tests to measure cognitive and motor functions. Participants may opt-in for research procedures such as phlebotomy, skin biopsy, leukapheresis, and lumbar puncture to obtain biospecimens for laboratory research, and magnetic resonance imaging or transcranial magnetic stimulation may be used to explore biomarkers of disease.

Outcome measures

Clinical information will be analyzed as part of our research to identify common features and differences among participants.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients will be included if they

* Are age 18 or older
* Have been given a diagnosis by a neurologist of frontotemporal dementia, primary progressive aphasia, semantic dementia, motor neuron disorder, amyotrophic lateral sclerosis, progressive bulbar palsy, corticobasal syndrome, Huntington disease or other related adult-onset neurodegenerative disorder OR
* Carry a mutation in a gene that causes familial ALS or FTD

EXCLUSION CRITERIA:

Patients will be excluded if they

* Have other major neurological or medical diseases that may cause progressive weakness or cognitive dysfunction, such as structural brain or spinal cord disease, metabolic diseases, paraneoplastic syndromes, infectious diseases, peripheral neuropathy or radiculopathy or other significant neurological abnormalities.
* Have an unstable medical condition that, in the opinion of the investigators, makes participation unsafe
* Require daytime ventilator support at the time of study entry
* Are unable to travel to NIH
* Patients with pacemakers or other implanted electrical devices, brain stimulators, dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pumps, or shrapnel fragments, metal fragments in the eye) will not be excluded but will not undergo magnetic resonance imaging.
* Patients with tattoos above the neck or permanent make up will be excluded from undergoing 7T MRI.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with a diagnosis of ALS, FTD, or a related adult-onset neurodegenerative disorder
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2017-10-11 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Clinical information | 10/30/2027
  Clinical information will be analyzed as part of our research to identify common features and differences among participants.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Y Kwan, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided.

REFERENCES:
- [Background] Snowden JS, Adams J, Harris J, Thompson JC, Rollinson S, Richardson A, Jones M, Neary D, Mann DM, Pickering-Brown S. Distinct clinical and pathological phenotypes in frontotemporal dementia associated with MAPT, PGRN and C9orf72 mutations. Amyotroph Lateral Scler Frontotemporal Degener. 2015;16(7-8):497-505. doi: 10.3109/21678421.2015.1074700. Epub 2015 Oct 16. PMID 26473392
- [Background] Renton AE, Majounie E, Waite A, Simon-Sanchez J, Rollinson S, Gibbs JR, Schymick JC, Laaksovirta H, van Swieten JC, Myllykangas L, Kalimo H, Paetau A, Abramzon Y, Remes AM, Kaganovich A, Scholz SW, Duckworth J, Ding J, Harmer DW, Hernandez DG, Johnson JO, Mok K, Ryten M, Trabzuni D, Guerreiro RJ, Orrell RW, Neal J, Murray A, Pearson J, Jansen IE, Sondervan D, Seelaar H, Blake D, Young K, Halliwell N, Callister JB, Toulson G, Richardson A, Gerhard A, Snowden J, Mann D, Neary D, Nalls MA, Peuralinna T, Jansson L, Isoviita VM, Kaivorinne AL, Holtta-Vuori M, Ikonen E, Sulkava R, Benatar M, Wuu J, Chio A, Restagno G, Borghero G, Sabatelli M; ITALSGEN Consortium; Heckerman D, Rogaeva E, Zinman L, Rothstein JD, Sendtner M, Drepper C, Eichler EE, Alkan C, Abdullaev Z, Pack SD, Dutra A, Pak E, Hardy J, Singleton A, Williams NM, Heutink P, Pickering-Brown S, Morris HR, Tienari PJ, Traynor BJ. A hexanucleotide repeat expansion in C9ORF72 is the cause of chromosome 9p21-linked ALS-FTD. Neuron. 2011 Oct 20;72(2):257-68. doi: 10.1016/j.neuron.2011.09.010. Epub 2011 Sep 21. PMID 21944779
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2017-N-0131.html